CLINICAL TRIAL: NCT04718545
Title: Treatment of Localized Gingival Recession Defects at Lower Mandibular Incisors Using a Modified-free Gingival Graft: a Randomized Clinical Trial
Brief Title: Effectiveness of Modified-free Gingival Graft for Treatment of Localized Gingival Recession Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OCarcuac-modFGG
Record Dates: First submitted 2021-01-16; First posted 2021-01-22 (Actual); Results first posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Gingival Recession, Localized
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free Gingival Graft (Active Comparator): A mucogingival surgery where a gingival graft harvested from the palate is placed on a conventionally prepared recipient site and sutured to cover the mucosal recession
  Interventions: Procedure: Mucogingival surgery
- Modified Free Gingival Graft (Experimental): A mucogingival surgery where a gingival graft harvested from the palate is placed on a modified recipient site and sutured to cover the mucosal recession
  Interventions: Procedure: Mucogingival surgery

INTERVENTIONS:
Procedure: Mucogingival surgery — The gingival recession at mandibular incisor site will be covered by a gingival graft harvested from the palate.

SUMMARY:
The aim of the present study is to evaluate, whether use of the modified free gingival graft (mod-FGG) technique improves treatment outcomes after surgical root coverage at mandibular incisors with gingival recession defects.

DETAILED DESCRIPTION:
Gingival recession defects (GRD), defined as displacement of the gingival margin apical to the cemento-enamel junction, are frequent clinical findings in the general population.

The major indications for root coverage procedures are improved esthetics, reduction of root hypersensitivity and the increase of the dimensions of keratinized tissue in order to facilitate infection control and prevent further progression of gingival recession defects. Numerous surgical techniques for root coverage have been suggested, with different degrees of success as assessed by the proportion of complete root coverage. The scientific evidence has revealed that mandibular incisors were associated with the least favourable outcomes when compared to other teeth. The lower success rate and lower predictability of root coverage procedures at lower incisors, teeth with the highest frequency of GRDs, may be related to the unfavorable anatomic conditions including marginal frenum attachment, high muscle pull and a shallow vestibule. These features are frequently encountered in the anterior area of the mandible, while they are rare in the maxillary anterior region.

The so-called "Free Gingival Graft" (FGG) was shown to be the most effective procedure for gingival augmentation at sites with minimal amount of keratinized tissue. Great variability in terms of proportion of root coverage (range: 11% to 87%; mean: 63%) has been reported when applying this technique, however. One of the challenges may be the inadequate blood supply to the portion of the FGG placed on the exposed root surface. A modified version of the FGG technique (mod-FGG) has been proposed, aiming to improve the vascularity of the recipient site over the denuded root surface. However, there is to date no scientific evidence whether the mod-FGG provides better clinical results than the conventional FGG.

The hypothesis of the study is that the mod-FGG will improve predictability and treatment outcomes for root coverage at mandibular incisors.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Periodontally and systemically healthy
* Full-mouth plaque score and full-mouth bleeding score ≤ 20% (measured at four sites per tooth)
* Thin phenotype
* Probing pocket depth (PPD) ≤3 mm
* Absence of excessive tooth mobility
* Absence of cervical composite restorations or non-carious cervical lesions
* Shallow vestibule

Exclusion Criteria:

* Pregnancy
* Smoking
* Alcoholism
* Para-functional habits
* Poor oral hygiene
* Excessive crowding or misalignment of teeth

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tord Berglundh, DDS, PhD, Study Chair — Goteborg University
Locations (1):
- Department of Periodontology, Institute of Odontology, Sahlgrenska Academy, University of Gothenburg, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tonetti MS, Jepsen S; Working Group 2 of the European Workshop on Periodontology. Clinical efficacy of periodontal plastic surgery procedures: consensus report of Group 2 of the 10th European Workshop on Periodontology. J Clin Periodontol. 2014 Apr;41 Suppl 15:S36-43. doi: 10.1111/jcpe.12219. PMID 24640999
- [Result] Cairo F. Periodontal plastic surgery of gingival recessions at single and multiple teeth. Periodontol 2000. 2017 Oct;75(1):296-316. doi: 10.1111/prd.12186. PMID 28758301
- [Result] Cortellini P, Bissada NF. Mucogingival conditions in the natural dentition: Narrative review, case definitions, and diagnostic considerations. J Periodontol. 2018 Jun;89 Suppl 1:S204-S213. doi: 10.1002/JPER.16-0671. PMID 29926948
- [Result] Zucchelli G, Marzadori M, Mounssif I, Mazzotti C, Stefanini M. Coronally advanced flap + connective tissue graft techniques for the treatment of deep gingival recession in the lower incisors. A controlled randomized clinical trial. J Clin Periodontol. 2014 Aug;41(8):806-13. doi: 10.1111/jcpe.12269. Epub 2014 Jun 5. PMID 24802283
- [Result] Holbrook T, Ochsenbein C. Complete coverage of the denuded root surface with a one-stage gingival graft. Int J Periodontics Restorative Dent. 1983;3(3):8-27. No abstract available. PMID 6358084
- [Result] Cairo F, Nieri M, Pagliaro U. Efficacy of periodontal plastic surgery procedures in the treatment of localized facial gingival recessions. A systematic review. J Clin Periodontol. 2014 Apr;41 Suppl 15:S44-62. doi: 10.1111/jcpe.12182. PMID 24641000

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Free Gingival Graft | Modified Free Gingival Graft
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Free Gingival Graft | Modified Free Gingival Graft | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (10.9) | 35.8 (10.0) | 36.2 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 9 | 6 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United Arab Emirates | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Mean Mid-facial Recession Coverage (mRC)
Description: mRC measured as a percentage
Time Frame: up to 1 year
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | Free Gingival Graft | Modified Free Gingival Graft
Number analyzed (Participants) | 15 | 15
percentage | 60.7 [56.0 to 65.3] | 91.8 [87.1 to 96.4]

2. Secondary Outcome: Keratinized Tissue (KT) Gain
Description: KT gain measured in mm
Time Frame: up to 1 year
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Free Gingival Graft | Modified Free Gingival Graft
Number analyzed (Participants) | 15 | 15
mm | 2.2 (0.9) | 4.2 (0.8)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Free Gingival Graft | Modified Free Gingival Graft
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/45/NCT04718545/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/45/NCT04718545/ICF_001.pdf